CLINICAL TRIAL: NCT01394835
Title: Safety and Efficacy of Inhaled Alpha-1 Antitrypsin in Preventing Bronchiolitis Obliterable Syndrome in Lung Transplant Recipients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Mordechai Kramer MD, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAT-02
Record Dates: First submitted 2011-07-05; First posted 2011-07-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Lung Transplantation; Bronchiolitis Obliterable Syndrome
Keywords: Patient after lung transplantation
MeSH Terms: interventions — alpha 1-Antitrypsin

ARMS (1):
- Alpha -1 Antitrypsin (Experimental)
  Interventions: Drug: Alpha -1 Antitrypsin; Drug: Alpha-1 Antitrypsin; Drug: AAT

INTERVENTIONS:
Drug: Alpha -1 Antitrypsin — Inhalation twice daily of 160mg
Drug: Alpha-1 Antitrypsin — Inhalation twice daily .Dosage 160mg
Drug: AAT — Inhalation twice daily' 160mg

SUMMARY:
Bronchiolitis obliterable syndrome (BOS) is the most common cause of death in long-term survivors after lung transplantation and refractory to most interventions. Many risk factor for BOS were identified in previous studies such as acute cellular rejection, lymphocytic bronchiolitis, cytomegalovirus (CMV) and non-CMV respiratory infections, injury to the allograft or airways, Primary graft dysfunction, HLA mismatching, and organizing pneumonia. (Belperio JA. et al.). Neutrophils and their released products may be involved in the development of BOS. Neutrophilia was repeatedly observed in the bronchoalveolar lavage fluid of patients after lung transplantation. In addition, infiltration of neutrophils into the bronchial epithelium has been detected in patients with higher degrees of active airway damage. Neutrophils are capable of causing severe damage to the lung tissue by releasing toxic proteases and reactive oxygen species if not counterbalanced by the antiprotease/ antioxidant screen of the lung. Based on this background, a causal relationship between neutrophilia and the development of BOS has been proposed. (Hirsch J. et al.) Detection of unopposed Neutrophile elastase (NE) activity in BAL appears to correlate with poor outcome due to refractory BOS. Unopposed NE in these subjects may not only serve as a marker of evolving graft dysfunction but also participate in damaging the airways of the allograft and inhibit adequate bacterial clearance. Prevention of neutrophil sequestration or inhibition of NE may prevent or attenuate airway damage and improve bacterial clearance mechanisms. (Nutley D et al.) These data demonstrate the importance of neutrophils and unopposed NE in the pathogenesis of BOS and call for new approach to prevent or modulate BOS targeting this mechanism.

AAT is the main inhibitor of neutrophil elastase in the lower airways and patients with AAT deficiency have low concentrations of the protein in this region of the lung. This explains the proteinase/antiproteinase theory of the development of emphysema in deficient patients in which the amount of elastase released in the lung exceeds the amount of AAT. The net result is persistence of elastase activity leading to lung destruction and the pathological changes of emphysema. (Abusriwil H. et al.) The administration of the AAT is to address proteinase/antiproteinase imbalance.

Administration of AAT will help to prevent further destruction of the lung architecture and reduce the inflammatory dysregulation that causes pulmonary dysfunction. It is expected that by attacking a specific and previously untreated key component part of the pathophysiological cycle of BOS, AAT therapy would decrease the prevalence of BOS in lung transplant recipients and prolong life expectancy of these patients.

ELIGIBILITY:
Inclusion Criteria:• Patients aged ≥18 years

* Signature of informed consent
* Lung transplant recipient in the past 6 months.
* Stable concomitant therapy >2 weeks prior to visit 1
* Non-tobacco user of any kind
* No significant abnormalities in serum hematology, serum chemistry to the Principal Investigator's judgment((Hg>8g/dL ,Creatinine<2mg/dl,Liver enzymes<3*ULN)
* Non-pregnant, non-lactating female subjects, whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator, or who are more than 5 years post-menopausal or surgically sterilized or whose way-of-life excludes sexual activity.
* Sexually active female subjects of child-bearing potential, as well as male subjects, must use a medically acceptable effective contraceptive method (for male - method such us condoms; for female - methods such as oral contraceptive medication used for at least two weeks before study start, or a combination of any two of the following: diaphragm, cervical cap, condom or spermicide), before study start and throughout the entire duration of the study.

Exclusion Criteria:• Diagnosis of BOS with according to Estenne M. et al.

* Hospitalization within 1 month before study entry, not due to an airway disease
* Severe liver cirrhosis with ascites
* Hypersplenism
* Grade III/IV esophageal varices;
* Active pulmonary exacerbation within the 4 weeks prior to screening
* History of massive hemoptysis: greater than 200 cc in a 24 hour period
* Pregnancy or breastfeeding
* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with patient treatment, assessment, or compliance with the protocol.
* Fever at the time of the start of first (day #1) inhalation (oral temperature >38ºC)
* Evidence of uncontrolled hypertension
* Pulse >120/min (prior to study drug administration)
* Any serious malignancy except for basal and squamous (scaly or plate-like) cell skin cancer within the previous 3 years prior to study start
* Receipt of exogenous AAT within the last 6 months
* Previous enrolment in this study (subject can not be enrolled twice into the study)
* Evidence of congestive heart failure or other clinically significant cardiovascular conditions: myocardial infarction during the last year, arrhythmia requiring drug treatment during the last year, uncontrolled hypertension
* Current smoker (someone who has smoked within 4 weeks prior to screening)
* Subjects with an additional clinically significant inter-current illness (beside lung disease) (e.g., cardiac, hepatic, renal, endocrine, respiratory, neurological, hematological, neoplastic, immunological and skeletal) that the investigator determines that it could interfere with the safety or other assessments of this study
* Any evidence of alcohol abuse or history of abuse of illegal and/or legally prescribed drugs such as barbiturates, benzodiazepines, amphetamines, cocaine, opioids, and cannabinoids
* Being a sexually active female of child-bearing age without adequate contraception
* Any other factor that, in the opinion of the investigator, would prevent the subject form complying with the requirements of the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Clinical diagnosis of BOS according to Estenne M. et al Treatment of lung transplant recipients to prevent BOS Clinical diagnosis of BOS according to Estenne M. et al. Adverse events and conc | 12 Month
  Adverse events and concomitant medication recording and follow up. Safety/tolerability parameters at baseline (Day #1) will be compared with values generated at the following visits every 6 weeks (+/- 10 days).
  At all visits, AEs and concomitant medications will be recorded. Additionally, the study coordinator will check occurrence of AE and concomitant medications by a telephone visit

SECONDARY OUTCOMES:
Change in lung function test | 12 month
  Change in lung function FEV%, FEV1, FVC Baseline (Day #1) values of FEV1 and FVC (and FEV%) will be compared to the following visits every 6 weeks (+/- 10 days).
  Incidence of Acute cellular rejection. Incidence of respiratory infection leading to antibiotics administration according to the decision of the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, M.D, Principal Investigator — Rabin Medical Center